CLINICAL TRIAL: NCT02221791
Title: Comparison of Pure Epicatechin and Cocoa on Markers of Vascular Function
Acronym: FLAVO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FLAVO2
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-08

CONDITIONS: Endothelial Dysfunction; Bioavailability
Keywords: Flavan-3-ol; Flavonoids; Epicatechin; Cocoa; Chocolate; Endothelial function; Bioavailability

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pure Epicatechin (Active Comparator): Participants will consume 100mg of epicatechin (capsule) + 70g white chocolate
  Interventions: Dietary Supplement: Pure Epicatechin
- High flavan-3-ol cocoa (Active Comparator): Participants will consume 70g high flavan-3-ol cocoa (100mg epicatechin) + placebo capsule
  Interventions: Dietary Supplement: High flavan-3-ol cocoa
- Placebo (Placebo Comparator): Participants will consume 70g white chocolate + placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pure Epicatechin — Participants will consume 100mg of epicatechin (capsule) + 70g white chocolate
  Arms: Pure Epicatechin
Dietary Supplement: High flavan-3-ol cocoa — Participants will consume 70g high flavan-3-ol cocoa (100mg epicatechin) + placebo capsule
  Arms: High flavan-3-ol cocoa
Dietary Supplement: Placebo — Participants will consume 70g white chocolate + placebo capsules
  Arms: Placebo

SUMMARY:
Intervention studies support a protective effect of flavonoid-rich foods such as chocolate and tea on cardiovascular disease risk. In a previous study we found that pure epicatechin improves markers of vascular function and insulin resistance although the results were less pronounced than the majority of chocolate intervention studies.

The food matrix of chocolate or other compounds present in chocolate could play a role in the bioavailability of flavonoids, resulting in these heightened improvements in vascular function.

In this study we aim to compare the acute effects of pure epicatechin and high-flavonoid chocolate on markers of vascular function.

DETAILED DESCRIPTION:
Twenty male participants between the ages of 40 and 80 will visit the university on three days, separated by a 2-week washout. During each visit the participants will, in random order, be allocated to one of the three interventions:

1. High flavan-3-ol chocolate (70g) plus placebo capsule;
2. White chocolate (70g) plus 100mg of epicatechin in capsule form;
3. White chocolate (70g) plus placebo capsule; Measurements of vascular function will be taken before, and 2 hours after consumption of the supplements. In order to determine flavonoid bioavailability, 24-hour urine samples will be collected and 7 blood samples will be taken over a period of 8 hours.

The primary study parameter is the percentage change in Flow-Mediated Dilation (FMD) as a result of a high-flavonoid cocoa or epicatechin challenge. Additional study parameters include plasma flavonoid and nitric oxide concentrations as well as pulse wave analysis parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years,
* BMI between > 20 and ≤ 30
* No reported current or previous metabolic diseases,
* No history of cardiovascular diseases,
* No history of renal, liver or thyroid diseases,
* No history of gastrointestinal diseases,
* No diagnosed diabetes mellitus,
* Fasting laboratory parameters within normal range as judged by the study physician: renal function (serum creatinine, ureum), liver function (ALAT, ASAT, GGT), serum glucose and HDL, LDL and total cholesterol.

Exclusion Criteria:

* Body mass index >30 or ≤20 kg/m2
* Usage of CVD medication (e.g. anti-hypertensive and/or lipid-modifying medication, non-steroidal anti-inflammatory drugs, acetylsalicylic acid), antibiotics, corticosteroids or opioids and not able or willing to stop taking them from at least 4 weeks prior to the study
* Taking nutritional supplements and unwilling to discontinue
* Reported dietary habits: medically prescribed diet, slimming diet
* Reported average alcohol consumption greater than or equal to 3 glasses/d
* Reported intense sporting activities > 10 h/w
* Weight loss or weight gain of 5 kg or more during the last 2 months
* Smokers
* Vegetarians
* Problems with consuming the supplements or following the study guidelines
* Recent blood donation (i.e. 1 month) prior to the study and/or planned donation during and shortly after the study period
* Not agreeing to be informed about unexpected and medically relevant personal test-results, or not agreeing that their general practitioner will be informed about these results
* Participation in another biomedical trial less than 2 months before the start of the study or at the same time
* No signed informed consent form
* Unable to comply with the study procedure (e.g. holidays, urine collection, blood sampling)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Endothelium-dependent flow-mediated dilation as a result of high flavan-3-ol cocoa or pure epicatechin consumption. | Baseline and 2 hours after consumption
  Change in arterial diameter as a result of 5 minute arterial occlusion (200mmHg). Arterial diameter will be measured by means of ultrasonography.

SECONDARY OUTCOMES:
Change in nitric oxide as a result of high flavan-3-ol cocoa or pure epicatechin consumption | Baseline and 1 hr, 2hr, 3hr, 4hr, 6hr and 8hr after consumption
  Plasma analysis of nitric oxide
Changes in arterial augmentation index as measured by Pulse Wave Analysis | Baseline and 2 hours after consumption
  Measured in triplicate using a SphygmoCor device at baseline and 2 hours after consumption
Bioavailability of plasma epicatechin metabolites | Baseline and 1hr, 2hr, 3hr, 4hr, 6hr and 8hr after consumption
  Plasma analysis of epicatechin metabolites will be measured up to 8 hours after consumption of high flavan-3-ol cocoa or pure epicatechin
Bioavailability of urine epicatechin metabolites | 24 hour urine samples
  Urinary epicatechin metabolites will be measured in 24-hour urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hollman, Dr, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- See also: Website for the study (in dutch) — http://voedingsonderzoek.wur.nl/flavo2